CLINICAL TRIAL: NCT04626245
Title: Mindfulness & Daily Experiences Study
Brief Title: Mindfulness & Mechanisms Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lifespan (Other)
Responsible Party: Principal Investigator, Margaret Bublitz, Senior Research Scientist, Lifespan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1679889-1
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Hypertension in Pregnancy
Keywords: mindfulness; pregnancy; blood pressure; ecological momentary assessment
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to a mindfulness training condition or treatment as usual.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness training (Experimental): Phone-delivered mindfulness training
  Interventions: Behavioral: Mindfulness training
- Treatment as usual (Other): Prenatal care
  Interventions: Behavioral: Mindfulness training

INTERVENTIONS:
Behavioral: Mindfulness training — Phone-delivered brief mindfulness training based on principles of MBSR

SUMMARY:
Hypertensive disorders of pregnancy (HDP) are the most common medical condition affecting pregnancy and a leading cause of maternal morbidity and mortality in the Unites States. HDP also increase lifetime cardiac disease risk in women and infants. Current interventions to prevent HDP are limited, and interventions that do not include medications are minimally effective at preventing HDP. Mindfulness interventions hold promise as a intervention to prevent HDP that does not require pregnant women to take medications. Past research shows that mindfulness interventions reduce blood pressure in adults with hypertension and pre-hypertension. However, past studies of mindfulness interventions for pregnant women have not allowed women at risk for HDP to participate. The preliminary study of prenatal mindfulness training for women at risk for HDP demonstrated benefit on maternal blood pressure and fetal growth. However, the mechanisms explaining effects of prenatal mindfulness training on risk for HDP are unknown. Building upon these promising preliminary findings, the proposed clinical trial will measure daily experiences of stress, physiological reactivity to stress, and interpersonal processes before and after prenatal mindfulness training. The investigators hypothesize that mindfulness training will impact these processes, which may lead to improved maternal cardiovascular parameters and reduced risk for HDP. N=150 pregnant women at risk for HDP will be randomized to an 8-week phone-delivered mindfulness intervention or usual care. For every participant, we will measure maternal cardiovascular parameters (24-hour blood pressure and uterine artery resistance values by ultrasound Doppler) before and after the 8-week period. All participants will complete surveys of daily experiences for 2 weeks before and after the 8-week period to evaluate mechanisms of mindfulness training on maternal cardiovascular parameters. Daily experiences will be measured using surveys delivered via smartphone-app, ambient audio sampling, and wearable wrist-worn biosensor monitoring (heart rate and heart rate variability).

DETAILED DESCRIPTION:
Hypertensive disorders of pregnancy (HDP) are the most common medical conditions in pregnancy and a leading cause of maternal morbidity and mortality in the United States. HDP are also associated with significant financial costs to the US healthcare system; $2.18 billion is spent on treatment of affected mothers and infants in the first year after delivery. Women exposed to HDP are at increased lifetime risk for cardiovascular disease, dementia, and all-cause mortality. Current interventions to prevent HDP are limited and do not target underlying mechanisms of disease. Mindfulness training (MT) holds tremendous promise as a mind-body intervention to prevent HDP. MT is effective at reducing blood pressure in non-pregnant patients with pre-hypertension and hypertension and has proven more effective at blood pressure reduction than other stress management interventions. Results from the pilot RCT were the first to indicate that prenatal phone-delivered MT is feasible and had a medium to large effect on cardiovascular parameters in women at risk for HDP. However, the mechanisms through which prenatal MT affects cardiovascular parameters are not yet understood.

MT teaches participants to "attend and respond in a non-judgmental way to ordinary, everyday experiences." Theory and available evidence indicate that MT elicits relaxation, decreases stress biomarkers and autonomic activation, and decreases loneliness --- dynamic processes that may serve as pathways to improved cardiovascular parameters in women at risk for HDP. The proposed RCT will harness subjective and objective ecological momentary assessment (EMA) methodologies (in vivo repeated assessments) in combination with wearable biosensor technology to capture rich epochs of ecologically-valid psychological, physiological, and interpersonal processes through which MT may lead to improved maternal cardiovascular parameters. Pregnant women at risk for HDP will be randomized to an 8-week phone-delivered MT intervention or usual care. For every participant, the research team will measure maternal cardiovascular parameters (24-hour blood pressure and uterine artery resistance values by ultrasound Doppler) before and after the RCT. All participants will complete EMA for 2 weeks 'bursts' before and after the RCT to evaluate mechanisms of MT on cardiovascular parameters. EMA will include smartphone-app based experience sampling of psychological processes; smartphone-app based ambient audio sampling (i.e. the Electronically Activated Recorder [EAR] method) and wearable wrist-worn biosensor monitoring of physiological responses (heart rate and heart rate variability) to everyday experiences. Results will provide new insights into 1) effects of MT on cardiovascular parameters in pregnancy, 2) pathophysiological mechanisms of HDP, and 3) targets for new HDP prevention strategies.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* English speaking
* less than 20 weeks' gestation at enrollment
* Blood pressure < 140/90
* Moderate to high risk for hypertensive disorders of pregnancy

Exclusion Criteria:

* Multiple gestations
* current severe depression or psychosis
* ongoing mind-body practice (e.g., yoga, meditation, mindfulness => once a week).

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Perceived stress and mood responses to momentary stress | Before and after the intervention, approximately 3 months
  Ecological momentary assessment surveys will query for maternal mood and perceived stress throughout the day.

SECONDARY OUTCOMES:
Heart rate response to momentary stress | Before and after the intervention, approximately 3 months
Perceived and received support in response to momentary stress | Before and after the intervention, approximately 3 months
  Ecological momentary assessment and audio recording will be used to measure perceived and received social support and loneliness throughout the day.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret H Bublitz, Principal Investigator — The Miriam Hospital
Locations (1):
- Women's Medicine Collaborative, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No